CLINICAL TRIAL: NCT01053195
Title: A Community-based Lifestyle Intervention to Reduce the Risk of Diabetes in Qingdao, China----Qingdao Diabetes Prevention Project (2005-2012)
Brief Title: Qingdao Diabetes Prevention Project
Acronym: QDDPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: The World Diabetes Foundation (Other); Qingdao Centers for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Qing Qiao, MD, Ph.D, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WDF07-308
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; prevention; intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): In the project areas, lifestyle counseling will be given every three months to individuals having prediabetes and every six months to those with normal glucose levels.
  Interventions: Behavioral: Lifestyle counseling
- Control (No Intervention): No intervention activity will be assigned for participants enrolled from the control areas.

INTERVENTIONS:
Behavioral: Lifestyle counseling — Non-diabetic high-risk subjects enrolled will be eligible for individual and/or group lifestyle counseling. The intervals of the counseling sessions depend on the glucose levels of the high-risk individuals, every three months for those having prediabetes and every six months for those with normal glucose levels but high risk score.
  Arms: Lifestyle counseling

SUMMARY:
Qingdao Diabetes Prevention Project aims to translate the trial experience to communities with specific objectives to:

* raise the public awareness of diabetes and diabetes risk factors
* promote healthy lifestyle of the entire targeting population
* reduce the number of people with obesity
* reduce the number of high-risk people developing diabetes through lifestyle intervention
* prevent the diabetic complications
* evaluate the effect and the cost of the community-based prevention project. The project is community-based targeting at the entire population of 1.94 million living in four administration districts of the city of Qingdao in China. In the first phase of the project (2005-2008) the work emphasis is on health promotion, training over 2000 primary care professionals and 300 school health nurses and establishing a network consisting of 600 community clinics. In the second phase (2008-2012) lifestyle counseling sessions will be provided to about 242112 high-risk individuals identified, and the efficacy and the cost of the project will be evaluated at the end of the project in 2012.

DETAILED DESCRIPTION:
The Qingdao Diabetes Prevention Project targets at two urban districts of Shinan and Shibei and two rural counties of Huangdao and Jiaonan, covering 1.94 million of people living in 512 urban communities and 1128 rural natural villages. There are 637000 households in the targeting districts.

In the first 3-years (2005-2008) we have focused on preparing educational materials, health promotion, distributing the project materials, training health professionals, establishing the project networks, identifying high-risk individuals etc., while from 2008-2011 we will transfer our working emphasis on lifestyle intervention to those with high-risk for diabetes.

According to the data collected in 2006, about 456288 individuals aged 35 years or older are estimated to have a risk score >=14. We estimate that at least 65% of the non-diabetic high-risk individuals (n=242112) will be identified and referred to one of the 600 community clinics for lifestyle counseling and intervention.

Lifestyle intervention includes individual and group counseling sessions organised by the community doctors in a real life setting. The intervals of the counseling sessions depend on the glucose levels of the high-risk individuals, every three months for those having impaired fasting glucose or/and impaired glucose tolerance and every six months for those with normal glucose levels but with high risk score. At the end of the project, the cost-effectiveness of the community-based intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* individuals Aged 35 years or older
* individuals at high risk for diabetes identified by a risk score assessment
* individuals with baseline measurement of glucose

Exclusion Criteria:

* individuals with a prior history of diabetes or taking antidiabetic drugs

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276793 (Actual)
Dates: Start 2005-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes | 7-8 years

SECONDARY OUTCOMES:
Cost-effectiveness of the lifestyle intervention | 7-8 years

CONTACTS AND LOCATIONS:
Overall Officials: Qing Qiao, MD, PhD, Principal Investigator — Department of Public Health, University of Helsinki
Locations (1):
- Qingdao Municipal Center for Disease Control & Prevention, Qingdao, Shandong, China

REFERENCES:
- [Background] Dong Y, Gao W, Nan H, Yu H, Li F, Duan W, Wang Y, Sun B, Qian R, Tuomilehto J, Qiao Q. Prevalence of Type 2 diabetes in urban and rural Chinese populations in Qingdao, China. Diabet Med. 2005 Oct;22(10):1427-33. doi: 10.1111/j.1464-5491.2005.01658.x. PMID 16176207
- [Background] Pan XR, Hu YH, Li GW, Liu PA, Bennett PH, Howard BV. Impaired glucose tolerance and its relationship to ECG-indicated coronary heart disease and risk factors among Chinese. Da Qing IGT and diabetes study. Diabetes Care. 1993 Jan;16(1):150-6. doi: 10.2337/diacare.16.1.150. PMID 8422770
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Jacobs-van der Bruggen MA, Bos G, Bemelmans WJ, Hoogenveen RT, Vijgen SM, Baan CA. Lifestyle interventions are cost-effective in people with different levels of diabetes risk: results from a modeling study. Diabetes Care. 2007 Jan;30(1):128-34. doi: 10.2337/dc06-0690. PMID 17192345
- [Background] Ning F, Pang ZC, Dong YH, Gao WG, Nan HR, Wang SJ, Zhang L, Ren J, Tuomilehto J, Hammar N, Malmberg K, Andersson SW, Qiao Q; Qingdao Diabetes Survey Group. Risk factors associated with the dramatic increase in the prevalence of diabetes in the adult Chinese population in Qingdao, China. Diabet Med. 2009 Sep;26(9):855-63. doi: 10.1111/j.1464-5491.2009.02791.x. PMID 19719705
- [Derived] Ning F, Zhao J, Zhang L, Wang W, Sun X, Song X, Zhang Y, Xin H, Gao W, Gao R, Zhang D, Pang Z. Famine exposure in early life and type 2 diabetes in adulthood: findings from prospective studies in China. Nutr Res Pract. 2023 Aug;17(4):780-788. doi: 10.4162/nrp.2023.17.4.780. Epub 2023 Mar 13. PMID 37529266